CLINICAL TRIAL: NCT07400198
Title: Identification of Gait-related Digital Biomarkers of Bone Health in Spinal Muscular Atrophy
Brief Title: Gait and Bone Health in SMA
Status: Recruiting | Type: Observational
Sponsor: Jacqueline Montes (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor-Investigator, Jacqueline Montes, Professor of Rehabilitation and Regenerative Medicine, Columbia University
Organization: Columbia University (Other)
Other Study IDs: AAAV3667
Record Dates: First submitted 2025-12-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Spinal Muscular Atrophy Type 3; Ambulatory Spinal Muscular Atrophy
Keywords: spinal muscular atrophy; SMA; instrumented insole; bone health; fracture; bone mineral density; gait; low bone mass
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood; Muscular Atrophy, Spinal; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood for assay of bone biomarkers: calcium serum, 25-hydroxyvitamin D2/D3 (vitamin D), bone-specific alkaline phosphatase, C-terminal telopeptide serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spinal Muscular Atrophy: Ambulatory children and adults at least 8 years old by the time of enrollment with genetically confirmed SMA.

SUMMARY:
The objective of this study is to understand how spatiotemporal and kinetic gait parameters are associated with bone health in pwSMA who are receiving DMT. We hypothesize that gait parameters are associated with BMD and can determine fracture risk in pwSMA. This is an observational study that involves one in-clinic visit (approximately 3 hours) with remote follow-up visits (approximately 15 minutes) every 3 months for 1 year to collect fracture and medical history. Each of the assessments included in this study are non-interventional and are not intended as a treatment nor are they at the level of standard of care.

DETAILED DESCRIPTION:
Addressing bone health is a high priority and remains a concern for the SMA community despite the availability of DMTs. Fractures often have devastating, irrecoverable impacts on function, especially in ambulatory pwSMA. While the most recent standards of care for SMA recommend annual screening, supportive treatments are not recommended until there has been a fracture, a reactive approach which may not be enough to mitigate LBM. Implementing novel, wearable technology and machine learning (ML) models to identify fracture risk will lead to a proactive approach to manage bone health and attenuate the negative sequalae of fractures. This is an observational cross-sectional study of ambulatory children and adults with SMA. The aims of this study are to (1) Identify gait-related digital biomarkers of bone health in ambulatory pwSMA, (2) Determine the ability of digital biomarkers to differentiate between pwSMA with and without a history of fractures, and (3) Investigate the ability of risk profiles derived from the digital biomarkers to predict prospective fractures over one year.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of 5qSMA
* Between 8 and 50 years of age
* Able to walk 10 meters without support or an assistive device
* All participants who meet the inclusion criteria regardless of treatment status will be included, including those on adjuvant therapies, whether investigational or approved

Exclusion Criteria:

* Injury or surgery within previous 3 months that would impact ability to perform in-clinic gait assessments
* Unwilling or unable to comply with all study procedures
* Age less than 8 or over 50 years

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study sample will include 22 ambulatory SMA participants.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Dual X-Ray Absorptiometry (DXA) | Baseline
  Bone mineral density (BMD), a measure of the mineral content in bones is assessed using dual x-ray absorptiometry (DXA). DXA can be used to identify individuals with low bone mass (LBM). DXA uses low-power x-ray and is a safe and reliable measure validated to diagnose osteoporosis. DXA provides a t-score and z-score so that based on age, low bone mass can be appropriately determined. DXA also provides a subtotal BMD score as well as scores specific to certain body regions, both of which will be utilized in the first aim.
Blood collection | Baseline
  Blood will be collected to assess for routine markers related to bone mineral density. Blood will be tested for levels of calcium, vitamin D, bone alkaline phosphatase (BALP), and C-terminal telopeptide of type I collagen (CTx). The amount of blood collected will be within hospital rules for children. The total amount of blood will be approximately 2 mL or 1/2 a teaspoon. BALP is a bone formation marker while CTx is a bone resorption marker. Calcium and vitamin D are known to be positively associated with BMD.
Fracture history | Baseline, months 3, 6, 9, and 12
  Details regarding lifetime fracture history will be collected via questioning at the in-clinic visit and during remote follow up visits, every three months for one year. The participant will be asked to describe each incident separately, including the age at fracture, mechanism of injury (how it happened, its nature, and force), any preceding events like falls or dizziness, and associated symptoms. Fractures will be characterized by location, type and treatment (surgical or conservative).
Fall history | Baseline, months 3, 6, 9 and 12
  Details regarding falls, that occurred within the past year, will be collected using a structured questionnaire at the in-clinic visit and during the one-year follow-up. Falls will be described by mechanism, environment and outcome.
Collection of spatiotempoal and kinetic gait parameters using instrumented insoles (AI-Sole) | Baseline
  Stride-by-stride spatiotemporal and kinetic gait parameters will be collected with AI-Sole continuously during the 6MWT. Spatiotemporal parameters included stride length (SL), stride velocity (SV), percent time in stance phase (%St), and percent time in terminal double support (%DS). Kinetic parameters included the anteroposterior (AP-COP) and mediolateral (ML-COP) ranges of the center-of-pressure normalized by shoe size, as well as the Absolute COP-Cyclogram Asymmetry Index (|ASI|).
Six Minute Walk Test | Baseline
  Participants will complete the six minute walk test in a corridor which includes the instrumented walkway, while wearing the insoles. This is to measure spatial parameters, kinetic parameters, temporal parameters, and metrics of cumulative activity in order to compare against the gold standard instrumented walkway. The six minute walk test is an objective evaluation of functional exercise capacity, and measures the maximum distance a person can walk in six minutes over a 25 meter course.
IPAQ-SF | Baseline
  A quantitative assessment of usual physical activity will be captured using the International Physical Activity Questionnaire Short Form (IPAQ-SF).The IPAQ-SF is a commonly used self-administered questionnaire designed to obtain internationally comparable data on health-related physical activity. The IPAQ-SF is composed of seven questions from four domains of physical activity, including vigorous and moderate physical activity, walking physical activity, and sitting time. A weighted total from vigorous physical activity, moderate physical activity, and walking physical activity is calculated to produce a total amount of physical activity in MET-min/week.

SECONDARY OUTCOMES:
Ten Meter Walk Run (10MWR) | Baseline
  The 10MWR is an objective evaluation of function that measures the speed at which an individual can complete 10 meters. Gait speed is a commonly used indicator in NMD, and this test can be done by either walking or running. The 10MWR has been demonstrated to be safe to administer in individuals with SMA.
Timed Up and Go Test (TUG) | Baseline
  The TUG test, a method to assess balance and mobility, measures the time it takes an individual to stand up from a chair, walk 3 meters, turn around, and sit down in the same chair. In SMA, TUG scores are associated with total leg and knee flexor strength, gross motor function, the 10-meter walk/run, and 6MWT. TUG test is a sensitive and reliable measure of functional impairment in inherited neuromuscular disorders.
30 Second Sit to Stand (30-STS) | Baseline
  The 30-STS test is used to evaluate basic muscle power and function. The participant is to complete as many sit-to-stands as possible, with or without using their hands for support, in 30 seconds.

OTHER OUTCOMES:
SMA EFFORT | Baseline
  The SMA EFFORT is a perceived physical fatigability patient-reported outcome measure (PROM) that provides a percent (PPF%) total score to each participant based on their participation over the past 30 days. PPF% total scores are calculated as the sum of activity item ratings divided by the number of items rated multiplied by five (highest rating on Likert scale), with higher scores indicating greater perceived physical fatigability (PPF).Participants are instructed to not endorse any item that has not been performed in the past 30 days, ensuring a PPF% total score that is unique to their current level of function. In addition to the PPF% total score (across all activities performed), PPF% subscale scores corresponding to the specific activities across 4 different domains of function are similarly derived (Exercise/Recreation, Mobility, Postural Control, and Activities of Daily Living (ADLs).

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided